CLINICAL TRIAL: NCT02255123
Title: A Retrospective Multicenter Study to Determine 4-Year Clinical Outcomes in Subjects Previously Enrolled in the CTOT-05 Study (CTOT-18)
Brief Title: Retrospective Multicenter Study to Determine 4-Year Clinical Outcomes in Subjects Previously Enrolled in the CTOT-05 Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOT-18
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a multicenter, non-randomized, retrospective study to collect long term (4 years post-transplant) clinical outcome data on subjects previously enrolled in the CTOT-05 study (NCT00466804) to evaluate participant and graft survival.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously enrolled in the CTOT-05 study
2. Subjects 4 years post-transplant (+/- 6 months).

Exclusion Criteria:

1. Withdrawal of consent from the CTOT-05 study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population was selected based on their previous participation in the parent study (CTOT-05). Participants enrolled in this study are at least 4 years post-transplant as of July 2014.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite incidence of Death, Re-transplantation or re-listed for transplantation, Coronary stent, Myocardial Infarction and Clinical evidence of CAV per ISHLT grading | 48 months (+/- 6 months) after primary transplantation
  Coronary Artery Vasculopathy (CAV)
  International Society for Heart and Lung Transplantation Registry (ISHLT)

SECONDARY OUTCOMES:
Incidence of death | 48 months (+/- 6 months) after primary transplantation
Incidence of re-transplantation or re-listed for transplantation | 48 months (+/- 6 months) after primary transplantation
Incidence of coronary stent | 48 months (+/- 6 months) after primary transplantation
Incidence of myocardial infarction | 48 months (+/- 6 months) after primary transplantation
Incidence of clinical evidence of CAV per ISHLT grading | 48 months (+/- 6 months) after primary transplantation
  Coronary Artery Vasculopathy (CAV)
  International Society for Heart and Lung Transplantation Registry (ISHLT)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Heeger, M.D., Study Chair — Icahn School of Medicine at Mount Sinai; Anil K. Chandraker, M.D., Study Chair — Brigham and Women's Hospital
Locations (12):
- United States (12):
  - University of California at San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Medical City Dallas Hospital/ CRSTI, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Starling RC, Stehlik J, Baran DA, Armstrong B, Stone JR, Ikle D, Morrison Y, Bridges ND, Putheti P, Strom TB, Bhasin M, Guleria I, Chandraker A, Sayegh M, Daly KP, Briscoe DM, Heeger PS; CTOT-05 consortium. Multicenter Analysis of Immune Biomarkers and Heart Transplant Outcomes: Results of the Clinical Trials in Organ Transplantation-05 Study. Am J Transplant. 2016 Jan;16(1):121-36. doi: 10.1111/ajt.13422. Epub 2015 Aug 10. PMID 26260101
- See also: The National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/